CLINICAL TRIAL: NCT05423743
Title: The INSPIRE-ASP Trial (INtelligent Stewardship Prompts to Improve Real-Time Empiric Antibiotic Selection for Patients) for Abdominal (ABD) Infections
Brief Title: INSPIRE Trial for Abdominal Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Hospital Corporation of America (Industry); University of California, Irvine (Other); University of Massachusetts, Amherst (Other); Brigham and Women's Hospital (Other); Rush University (Other)
Responsible Party: Principal Investigator, Richard Platt, MD, MSc, Professor and Chair, Department of Population Medicine, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PH000763B_ABD
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Abdominal (ABD) Infection
Keywords: ABD; CPOE; Empiric Therapy
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: This cluster-randomized trial will assess a novel quality improvement antibiotic stewardship strategy for empiric antibiotic selection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Routine Care (Active Comparator): Continuation of routine antibiotic stewardship strategies.
  Interventions: Other: Arm 1: Routine Care
- Arm 2: INSPIRE Stewardship Bundle (Active Comparator): Use of computerized physician order entry (CPOE) smart prompts, clinician feedback, and activities to support CPOE adoption (including education and alignment of CPOE workflows) to guide empiric choice of antibiotics for abdominal infection in the first 3 days of hospitalization.
  Interventions: Other: Arm 2: INSPIRE Stewardship Bundle for Abdominal Infection

INTERVENTIONS:
Other: Arm 1: Routine Care — Routine Antibiotic Stewardship Arm - Continuation of antibiotic stewardship activities in accordance with national standards.
  Arms: Arm 1: Routine Care
Other: Arm 2: INSPIRE Stewardship Bundle for Abdominal Infection — Quality improvement intervention that includes (1) computerized physician order entry (CPOE) decision support alert that provides physicians with patient-specific risk estimates for having an abdominal infection due to a multidrug-resistant organism (MDRO) and recommends standard spectrum antibiotics for low risk patients in the first 3 days of hospitalization; (2) clinician feedback reports, and (3) activities to support CPOE adoption (including education and alignment of CPOE workflows). Other antibiotic stewardship activities to continue in accordance with national standards.
  Arms: Arm 2: INSPIRE Stewardship Bundle

SUMMARY:
The INSPIRE Abdominal Infection Trial is a cluster-randomized controlled trial of HCA Healthcare hospitals comparing routine empiric antibiotic stewardship practices with real-time, precision medicine computerized physician order entry (CPOE) smart prompts providing the probability that a non-critically ill adult admitted with abdominal infection is infected with a resistant pathogen.

Note: enrolled "subjects" represent 102 individual HCA Healthcare hospitals that have been randomized into 92 clusters. Hospitals were grouped into the same randomization cluster if they shared campuses or antibiotic stewardship staff.

ELIGIBILITY:
Facility Inclusion Criteria:

1. HCA Healthcare hospitals admitting adults for abdominal infection
2. Facility use of MEDITECH as their electronic health record system

Facility Exclusion Criteria:

-

Note: unit of randomization is the hospital, however the computerized physician order entry (CPOE) alert intervention will calculate risk estimates for adults age >=18 admitted to non-intensive care unit wards and who are ordered to receive extended-spectrum antibiotics for abdominal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198480 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Gohil, MD, MPH, Study Director — UC Irvine Division of Infectious Diseases; Susan Huang, MD, MPH, Principal Investigator — UC Irvine Division of Infectious Diseases; Richard Platt, MD, MS, Principal Investigator — Harvard Pilgrim Health Care Institute/Harvard Medical School
Locations (101):
- United States (101):
  - Riverside Community Hospital, Riverside, California
  - Regional Medical Center of San Jose, San Jose, California
  - Good Samaritan Hospital, San Jose, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - West Hills Hospital & Medical Center, West Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Blake Medical Center, Bradenton, Florida
  - Brandon Regional Hospital, Brandon, Florida
  - Oak Hill Hospital, Brooksville, Florida
  - Englewood Community Hospital, Englewood, Florida
  - Fort Walton Beach Medical Center, Fort Walton Beach, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Regional Medical Center of Bayonet Point, Hudson, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Lake City Medical Center, Lake City, Florida
  - Largo Medical Center, Largo, Florida
  - Northwest Medical Center, Margate, Florida
  - Mercy Hospital, Miami, Florida
  - Kendall Regional Medical Center, Miami, Florida
  - Orange Park Medical Center, Orange Park, Florida
  - Oviedo Medical Center, Oviedo, Florida
  - Gulf Coast Regional Medical Center, Panama City, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - St. Lucie Medical Center, Port Saint Lucie, Florida
  - Doctors Hospital of Sarasota, Sarasota, Florida
  - Palms of Pasadena, St. Petersburg, Florida
  - Northside Hospital, St. Petersburg, Florida
  - St. Petersburg General Hospital, St. Petersburg, Florida
  - South Bay Hospital, Sun City Center, Florida
  - Capital Regional Medical Center, Tallahassee, Florida
  - HCA Florida South Tampa Hospital, Tampa, Florida
  - HCA Florida West Tampa Hospital, Tampa, Florida
  - Medical Center of Trinity, Trinity, Florida
  - JFK Medical Center - North Campus, West Palm Beach, Florida
  - Fairview Park Hospital, Dublin, Georgia
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Menorah Medical Center, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wesley Woodlawn Hospital & ER, Wichita, Kansas
  - TriStar Greenview Regional Hospital, Bowling Green, Kentucky
  - Lakeview Regional Medical Center, Covington, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Lee's Summit Medical Center, Lee's Summit, Missouri
  - Southern Hills Hospital & Medical Center, Las Vegas, Nevada
  - Sunrise Hospital & Medical Center, Las Vegas, Nevada
  - Trident Medical Center, Charleston, South Carolina
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Parkridge East Hospital, Chattanooga, Tennessee
  - TriStar Horizon Medical Center, Dickson, Tennessee
  - TriStar Hendersonville Medical Center, Hendersonville, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - TriStar Southern Hills Medical Center, Nashville, Tennessee
  - TriStar StoneCrest Medical Center, Smyrna, Tennessee
  - Medical City Arlington, Arlington, Texas
  - St. David's Medical Center, Austin, Texas
  - St. David's North Austin Medical Center, Austin, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - HCA Houston Healthcare Conroe, Conroe, Texas
  - Corpus Christi Medical Center - Bay Area, Corpus Christi, Texas
  - Corpus Christi Medical Center - Doctors Regional, Corpus Christi, Texas
  - Corpus Christi Medical Center - Heart Hospital, Corpus Christi, Texas
  - Medical City Dallas, Dallas, Texas
  - Medical City Denton, Denton, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - Del Sol Medical Center, El Paso, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - Medical City Alliance, Fort Worth, Texas
  - Medical City Frisco, Frisco, Texas
  - HCA Houston Healthcare West, Houston, Texas
  - Medical City Las Colinas, Irving, Texas
  - HCA Houston Healthcare Kingwood, Kingwood, Texas
  - Medical City Lewisville, Lewisville, Texas
  - Methodist Hospital Northeast, Live Oak, Texas
  - Rio Grande Regional Hospital Main Campus, McAllen, Texas
  - Medical City McKinney, McKinney, Texas
  - Medical City North Hills, North Richland Hills, Texas
  - HCA Houston Healthcare Southeast, Pasadena, Texas
  - HCA Houston Healthcare Pearland, Pearland, Texas
  - Medical City Plano, Plano, Texas
  - St. David's Round Rock Medical Center, Round Rock, Texas
  - Methodist Hospital Texsan, San Antonio, Texas
  - Methodist Hospital Metropolitan, San Antonio, Texas
  - Methodist Hospital | Specialty and Transplant, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - HCA Houston Healthcare Mainland, Texas City, Texas
  - Medical City Weatherford, Weatherford, Texas
  - HCA Houston Healthcare Clear Lake, Webster, Texas
  - Ogden Regional Medical Center, Ogden, Utah
  - LewisGale Hospital Montgomery, Blacksburg, Virginia
  - LewisGale Hospital Pulaski, Pulaski, Virginia
  - Reston Hospital Center, Reston, Virginia
  - CJW Medical Center (Chippenham & Johnston Willis Campuses), Richmond, Virginia
  - Henrico Doctors' Hospital, Richmond, Virginia
  - LewisGale Medical Center, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gohil SK, Septimus E, Kleinman K, Varma N, Sands KE, Avery TR, Mauricio A, Sljivo S, Rahm R, Roemer K, Cooper WS, McLean LE, Nickolay NG, Poland RE, Weinstein RA, Fakhry SM, Guy J, Moody J, Coady MH, Smith KN, Meador B, Froman A, Eibensteiner K, Hayden MK, Kubiak DW, Burks C, Burgess LH, Calderwood MS, Perlin JB, Platt R, Huang SS. Improving Empiric Antibiotic Selection for Patients Hospitalized With Abdominal Infection: The INSPIRE 4 Cluster Randomized Clinical Trial. JAMA Surg. 2025 Jul 1;160(7):733-743. doi: 10.1001/jamasurg.2025.1108. PMID 40208583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 92 out of 142 HCA Healthcare hospitals were recruited for this trial. There was a 12-month baseline period (January 1, 2019-December 31, 2019), 5-month phase-in (August 2, 2022-December 31, 2022), and 12-month intervention (January 1, 2023-December 31,2023). Data from the phase-in period were excluded from all analyses (i.e., Baseline, Intervention, Outcome Measures, and Adverse Events).
Pre-assignment Details: 198,480 patients across 92 hospitals were randomized to either the routine stewardship group (Arm 1) or to the CPOE bundle (Arm 2); 2 hospitals were excluded because they divested from HCA Healthcare before the intervention period began.
Units Other Than Participants: Hospitals
Groups:
- Arm 1: Routine Stewardship: Continuation of routine antibiotic stewardship strategies.
  Arm 1: Routine Care: Routine Antibiotic Stewardship Arm - Continuation of antibiotic stewardship activities in accordance with national standards.
- Arm 2: INSPIRE CPOE Bundle: Use of computerized physician order entry (CPOE) smart prompts, clinician feedback, and activities to support CPOE adoption (including education and alignment of CPOE workflows) to guide empiric choice of antibiotics for abdominal infection in the first 3 days of hospitalization.
  Arm 2: INSPIRE Stewardship Bundle for Abdominal Infection: Quality improvement intervention that includes (1) computerized physician order entry (CPOE) decision support alert that provides physicians with patient-specific risk estimates for having an abdominal infection due to a multidrug-resistant organism (MDRO) and recommends standard spectrum antibiotics for low risk patients in the first 3 days of hospitalization; (2) clinician feedback reports, and (3) activities to support CPOE adoption (including education and alignment of CPOE workflows). Other antibiotic stewardship activities to continue in accordance with national standards.
Period: Baseline (12 Months)
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle
Started | 46725; 46 Hospitals | 46751; 46 Hospitals
Completed | 46725; 46 Hospitals | 46751; 46 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Intervention (12 Months)
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle
Started | 54384; 46 Hospitals | 50620; 44 Hospitals (2 hospitals were excluded from Arm 2: CPOE Bundle because they divested from HCA Healthcare before the intervention period began)
Completed | 54384; 46 Hospitals | 50620; 44 Hospitals (2 hospitals were excluded from Arm 2: CPOE Bundle because they divested from HCA Healthcare before the intervention period began)
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Population: Overall number of participants reflects the total across baseline and intervention periods.
  198,480 patients from 92 hospitals were randomized to a study group; Prior to the to start of the intervention period, 2 hospitals divested from the participating healthcare system, and thus were excluded from Arm 2: CPOE Bundle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle | Total
Number analyzed (Participants) | 101109 | 97371 | 198480
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  years
    Baseline (12 months): number analyzed (Participants) | 46725 | 46751 | 93476
    Baseline (12 months) | 61 (19) | 59 (19) | 60 (19)
    Intervention (12 months): number analyzed (Participants) | 54384 | 50620 | 105004
    Intervention (12 months) | 61 (19) | 59 (19) | 60 (19)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    Baseline (12 months): number analyzed (Participants) | 46725 | 46751 | 93476
    Baseline (12 months): Female | 28375 | 28249 | 56624
    Baseline (12 months): Male | 18185 | 18349 | 36534
    Baseline (12 months): Unknown | 165 | 153 | 318
    Intervention (12 months): number analyzed (Participants) | 54384 | 50620 | 105004
    Intervention (12 months): Female | 32114 | 29985 | 62099
    Intervention (12 months): Male | 22268 | 20635 | 42903
    Intervention (12 months): Unknown | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    Baseline (12 months): number analyzed (Participants) | 46725 | 46751 | 93476
    Baseline (12 months): Black | 4591 | 5754 | 10345
    Baseline (12 months): White | 35197 | 33004 | 68201
    Baseline (12 months): Other | 2915 | 1702 | 4617
    Baseline (12 months): Unknown | 4022 | 6291 | 10313
    Intervention (12 months): number analyzed (Participants) | 54384 | 50620 | 105004
    Intervention (12 months): Black | 5730 | 6033 | 11763
    Intervention (12 months): White | 39497 | 35429 | 74926
    Intervention (12 months): Other | 1981 | 1066 | 3047
    Intervention (12 months): Unknown | 7176 | 8092 | 15268

OUTCOME MEASURES:

1. Primary Outcome: Extended-Spectrum Days of Antibacterial Therapy (ES-DOT) Per Empiric Day
Description: Days-of-Therapy is a standardized national measure for antibacterial use in hospitals that counts each different antibiotic administered on each calendar day as one day of therapy, regardless of doses given.
  Extended-spectrum days-of-therapy per empiric day is defined as the summed number of different extended-spectrum antibiotics received per patient each calendar day, beginning at admission. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
  For example, 2 different extended-spectrum antibiotics administered at least once during each of the first 3 days would yield 6 days of extended-spectrum days-of-therapy.
Time Frame: First 3 calendar days of hospitalization for each patient during the 12-month baseline and 12-month intervention periods
Population: The total number of participants analyzed reported here is from the baseline and intervention periods
Measure: Number; unit: Extended-Spectrum Days-of-Therapy
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle
Number analyzed (Participants) | 101109 | 97371
Extended-Spectrum Days-of-Therapy
  Baseline (12 months): number analyzed (Participants) | 46725 | 46751
  Baseline (12 months) | 68616 | 68679
  Intervention (12 months): number analyzed (Participants) | 54384 | 50620
  Intervention (12 months) | 76605 | 50001

2. Secondary Outcome: Vancomycin Days of Antibacterial Therapy Per Empiric Day
Description: Days-of-Therapy is a standardized national measure for antibacterial use in hospitals that counts each different antibiotic administered on each calendar day as one day of therapy, regardless of doses given.
  Vancomycin days-of-therapy per empiric day is defined as the the number of days that vancomycin is received by a patient, averaged over the empiric period, and summed across all participants. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
Time Frame: as for outcome 1
Population: The total number of participants analyzed reported here is from the baseline and intervention periods
Measure: Number; unit: Vancomycin Days-of-Therapy
Arm/Group | Arm 1: Routine Care | Arm 2: INSPIRE Stewardship Bundle
Number analyzed (Participants) | 101109 | 97371
Vancomycin Days-of-Therapy
  Baseline (12 months): number analyzed (Participants) | 46725 | 46751
  Baseline (12 months) | 13019 | 13198
  Intervention (12 months): number analyzed (Participants) | 54384 | 50620
  Intervention (12 months) | 12780 | 13019

3. Secondary Outcome: Antipseudomonal Antibiotic Days Of Therapy (ES-DOT) Per Empiric Day
Description: Days-of-Therapy is a standardized national measure for antibacterial use in hospitals that counts each different antibiotic administered on each calendar day as one day of therapy, regardless of doses given.
  Antipseudomonal days-of-therapy per empiric day is defined as the summed number of different antipseudomonal antibiotics received per patient each calendar day, beginning at admission. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
  For example, 2 different antipseudomonal antibiotics administered at least once during each of the first 3 days would yield 6 days of antipseudomonal days-of-therapy.
Time Frame: as for outcome 1
Population: The total number of participants analyzed reported here is from the baseline and intervention periods
Measure: Number; unit: Antipseudomonal Days-of-Therapy
Arm/Group | Arm 1: Routine Care | Arm 2: INSPIRE CPOE Bundle
Number analyzed (Participants) | 101109 | 97371
Antipseudomonal Days-of-Therapy
  Baseline (12 months): number analyzed (Participants) | 46725 | 46751
  Baseline (12 months) | 49377 | 49249
  Intervention (12 months): number analyzed (Participants) | 54384 | 50620
  Intervention (12 months) | 56465 | 34362

4. Other Pre Specified Outcome: Intensive Care Unit (ICU) Transfer [Safety Outcome 1]
Description: Days from hospital admission until transfer to ICU, if that occurs. If it doesn't occur, the number of days is censored (capped) at the patient's hospital discharge or at the end of data collection. Almost all patients will be discharged before the end of trial data collection.
Time Frame: Duration of hospitalization for each patient during 12-month baseline and 12-month intervention periods
Population: The mean number of days to event here is from the the baseline and intervention periods
Measure: Mean (Standard Deviation); unit: Days to event
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle
Number analyzed (Participants) | 101109 | 97371
Days to event
  Baseline (12 months): number analyzed (Participants) | 46725 | 46751
  Baseline (12 months) | 5.4 (3.4) | 5.4 (3.4)
  Intervention (12 months): number analyzed (Participants) | 54384 | 50620
  Intervention (12 months) | 5.5 (3.5) | 5.5 (3.5)

5. Other Pre Specified Outcome: Length-of-stay [Safety Outcome 2]
Description: Days from hospital admission until discharge. If the patient remains in the hospital at the end of the trial data collection, the number of days is censored (capped) at that time. Almost all patients will be discharged before the end of trial data collection.
Time Frame: Duration of hospitalization for each patient during 12-month baseline and 12-month intervention periods
Population: The mean number of days to event here is from the baseline and intervention periods
Measure: Mean (Standard Deviation); unit: Days to event
Arm/Group | Arm 1: Routine Care | Arm 2: INSPIRE CPOE Bundle
Number analyzed (Participants) | 101109 | 97371
Days to event
  Baseline (12 months): number analyzed (Participants) | 46725 | 46751
  Baseline (12 months) | 5.5 (2.8) | 5.6 (2.9)
  Intervention (12 months): number analyzed (Participants) | 54384 | 50620
  Intervention (12 months) | 5.7 (2.9) | 5.8 (3.0)

6. Other Pre Specified Outcome: Extended-Spectrum Days of Therapy With Inpatient Extended-Spectrum (ES) Antibiotic Treatment After Empiric Period
Description: The number of different ES antibiotics received each day, on hospital days ≥4 and ≤14.
  Note: this outcome is intended for a secondary manuscript
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

7. Other Pre Specified Outcome: Empiric and Total Antibiotic Costs
Description: Empiric and total antibiotic costs for abdominal infection during hospitalization.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

8. Other Pre Specified Outcome: Incidence of Hospital-Onset C. Difficile
Description: Hospital-onset C. difficile positive tests (specimen obtained) on hospital days ≥4 and ≤14.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

9. Other Pre Specified Outcome: Incidence of Hospital-Onset MDRO-Positive Cultures
Description: Newly-detected hospital-onset MDRO-positive cultures on hospital days ≥4 and ≤14. Includes total MDRO and specific MDRO subsets.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: 12 months (baseline), 12 months (intervention)
Arm/Group | Arm 1: Routine Stewardship | Arm 2: INSPIRE CPOE Bundle
All-Cause Mortality (participants affected / at risk) | 0/101109 | 0/97371
Serious Adverse Events (participants affected / at risk) | 0/101109 | 0/97371
Other Adverse Events (participants affected / at risk) | 0/101109 | 0/97371

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05423743/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT05423743/SAP_001.pdf